CLINICAL TRIAL: NCT00079924
Title: Effects of Teriparatide in Postmenopausal Women With Osteoporosis Previously Treated With Alendronate or Raloxifene
Brief Title: Effects of Teriparatide in Postmenopausal Women With Osteoporosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 8141; B3D-MC-GHCM
Record Dates: First submitted 2004-03-18; First posted 2004-03-19 (Estimated); Last update posted 2007-05-25 (Estimated); Status verified 2007-05

CONDITIONS: Postmenopausal Osteoporosis
MeSH Terms: conditions — Osteoporosis, Postmenopausal | interventions — Teriparatide; Raloxifene Hydrochloride

INTERVENTIONS:
Drug: teriparatide
Drug: aldrenodate
Drug: raloxifene

SUMMARY:
Effects of Teriparatide in Postmenopausal Women Previously Treated with Alendronate or Raloxifene.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women aged at least 50 years
* A previous clinical diagnosis of osteoporosis
* At high risk for fracture
* Current therapy for at least 18 months prior to study entry with either raloxifene HCl or alendronate Na

Exclusion Criteria:

* History of metabolic bone disease other than osteoporosis
* History of malignant neoplasm within the last 5 years except for superficial basal cell carcinoma or squamous cell carcinoma

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200
Dates: Start 2004-11; Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Change in calcium values after beginning teriparatide

SECONDARY OUTCOMES:
Frequency of hypercalcemia, various calcium assessments, change in bone mineral density and tests of bone formation and resorption

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (10):
- United States (10):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM - 5PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Birmingham, Alabama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM - 5PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Huntsville, Alabama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM - 5PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Scottsdale, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM - 5PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jacksonville, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM - 5PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gainesville, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM - 5PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Des Moines, Iowa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM - 5PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rochester, Minnesota
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM - 5PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., West Haverstraw, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM - 5PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Charlotte, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM - 5PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tulsa, Oklahoma

REFERENCES:
- [Derived] Cosman F, Wermers RA, Recknor C, Mauck KF, Xie L, Glass EV, Krege JH. Effects of teriparatide in postmenopausal women with osteoporosis on prior alendronate or raloxifene: differences between stopping and continuing the antiresorptive agent. J Clin Endocrinol Metab. 2009 Oct;94(10):3772-80. doi: 10.1210/jc.2008-2719. Epub 2009 Jul 7. PMID 19584192
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com